CLINICAL TRIAL: NCT02844920
Title: Evaluation of Uterine Patency Following Sonography-guided Transcervical Ablation of Fibroids
Acronym: OPEN
Status: Completed | Type: Observational
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Other Study IDs: CL04897
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Uterine Fibroids; Adhesions
MeSH Terms: conditions — Leiomyoma; Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Fibroid Treatment: Intrauterine ultrasound guided radio-frequency ablation
  Interventions: Device: Intrauterine ultrasound guided radio-frequency ablation

INTERVENTIONS:
Device: Intrauterine ultrasound guided radio-frequency ablation — Radiofrequency ablation for the treatment of uterine fibroids
  Other Names: Sonata System

SUMMARY:
This study is designed to observe the presence or absence of intrauterine adhesions at 6 weeks after treatment with the Sonata® System through hysteroscopic evaluation by third party readers.

DETAILED DESCRIPTION:
Patients who agree to participate in this observational trial will have selected fibroid treatment with the Sonata System. Research participants will undergo hysteroscopy at 6 weeks following treatment to evaluate presence or absence of intrauterine adhesions.

Research participants will be asked to complete a quality of life questionnaire prior to and 6 weeks following treatment. Research participants will also complete a satisfaction survey and a diary that tracks their return to normal daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Have selected Sonata for treatment of fibroids in the presence of heavy menstrual bleeding
* Presence of at least one submucous myoma (type 1, type 2) or transmural fibroid (type 2-5)
* Willing and able to read, understand, and sign the informed consent form and to adhere to all study follow-up requirements

Exclusion Criteria:

* Preexisting adhesions within the endometrial cavity as indicated by an ESH score ≥ I as determined by the investigator
* One or more Type 0 fibroids and/or endometrial polyps of any size
* Any reason for which, in the opinion of the Investigator, the individual study patient is not appropriate or suitable for participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who desire treatment of intrauterine fibroids with RF ablation via the Sonata System.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (3):
  - Klinikum Mannheim Universitäts- Frauenklinik Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Klinikum Oldenburg, Oldenburg
  - Universitätsklinikum Tübingen, Tübingen
- Maxima Medisch Centrum (MMC), Veldhoven, Netherlands
- Universitätsklinik für Frauenheilkunde Inselspital Bern, Bern, Switzerland
- St. Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This observational study is intended to view the group as an entirety, individual participant data will be analyzed for adhesions but will not be shared independently.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fibroid Treatment
Started | 37
Completed Without Evaluable Videos | 1 (Participants with completed the follow-up but without evaluable hysteroscopy videos)
Completed With Evaluable Videos | 34 (Participants with completed the follow-up and evaluable hysteroscopy videos)
Completed, Eval. Data, Opposing Fibroids | 6 (Participants with completed the follow-up, evaluable hysteroscopy videos, and opposing fibroids)
Completed | 35 (Participants with completed the follow-up)
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Fibroid Treatment: Intrauterine ultrasound guided radio-frequency ablation Intrauterine ultrasound guided radio-frequency ablation: Radiofrequency ablation for the treatment of uterine fibroids
Arm/Group | Fibroid Treatment
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (5.23)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Newly Formed Intrauterine Adhesions Following RF Ablation of Fibroids
Description: Hysteroscopic evaluation by independent readers to determine the presence or absence of adhesions following transcervical RF ablation of fibroids with the Sonata system in participants who completed the follow-up assessment AND evaluable hysteroscopy videos.
Time Frame: 6 weeks
Population: Participants with completed follow-up assessment and had evaluable hysteroscopy videos.
Measure: Count of Participants; unit: Participants
Arm/Group | Fibroid Treatment
Number analyzed (Participants) | 34
Participants | 34

2. Secondary Outcome: Umber of Participants With Absence of Newly Formed Adhesions Following RF Ablation of Fibroids in Participants With Apposing Fibroids Treated
Description: As the risk of adhesion formation is higher when apposing fibroids are treated, this outcome measure assesses adhesiogenesis in the subgroup of the population who completed the follow-up assessment, had evaluable hysteroscopy videos, and had apposing fibroids treated.
Time Frame: 6 weeks
Population: Participants who completed the follow-up assessment, had evaluable hysteroscopy videos, and had apposing fibroids treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Fibroid Treatment
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Fibroid Treatment
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibroid Treatment (N=37)
Gall Stones (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT02844920/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT02844920/SAP_001.pdf